CLINICAL TRIAL: NCT07201376
Title: Tissue Oxygen Imager
Brief Title: Assessment of Skin Lesions Using a Tissue Oxygen Imager Based on Protoporphyrin IX (PPIX) Fluorescence. This is an Open-label, Non-randomized, Feasibility Study That Includes a One-time Application of an FDA Approved Medication Followed by Local Imaging for Benign Skin Growth and Lesions Clinically
Acronym: PPIX
Status: Recruiting | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Dartmouth College (Other)
Responsible Party: Principal Investigator, Michael S. Chapman, Principal Investigator, Dartmouth-Hitchcock Medical Center
Other Study IDs: STUDY02002181
Record Dates: First submitted 2025-09-19; First posted 2025-10-01 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-09

CONDITIONS: Non-Melanoma Skin Cancer (NMSC); Benign Skin Growth
Keywords: Benign Skin Growth; Non-Melanoma Skin Cancer
MeSH Terms: interventions — Aminolevulinic Acid; Gels

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Ameluz 10% Topical Gel — One-time topical application of 10% Ameluz gel for up to 1 hour
Device: Protoporphyrin IX — Tissue oxygen imaging using protoporphyrin IX (PIX), a non-significant risk device.

SUMMARY:
The primary objective of this study is the evaluation of the efficacy of the tissue oxygen imager based on PpIX DF in differentiating benign skin growth from non-melanoma skin cancer (NMSC).

DETAILED DESCRIPTION:
The present study is an open-label, non-randomized, feasibility study aiming to evaluate the ability of a non-significant risk tissue oxygen imager based on protoporphyrin IX (PpIX) delayed fluorescence (DF) for differentiating benign from malignant skin lesions and assessing tumor margins during Mohs micrographic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age.
* Histologic proof of non-melanoma skin cancer. Patients with different skin tones based on the Fitzpatrick Scale, who present with skin growth or lesions and are scheduled for resection.
* As determined by the enrolling physician or study team member, the patient must have the willingness and ability to understand and comply with study procedures.
* Women of childbearing potential (WOCBP): Premenopausal females who had at least one menstrual cycle in the past 12-months and capable to become pregnant, must have a negative serum beta-HCG pregnancy test result within seven days prior to start of study.
* Lesions must measure between 5 mm and 3 cm in diameter.

Exclusion Criteria:

* Patients who are <18 years of age
* Adults who are unable to provide informed consent.
* Known allergy to Ameluz
* Photosensitivity or photodermatoses or similar conditions.
* Patients with any serious underlying medical condition that would impair their ability to receive or tolerate the planned treatment and/or comply with study protocol, in the opinion of the investigator
* Known hypersensitivity to porphyrins or to any component of Ameluz, including soya bean phosphatidylcholine.
* Females who are currently breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be enrolled from the Dermatology Clinic where the study is being performed.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Detecting cutaneous malignant lesions using a non-invasive technique | Six months after the first enrollment
  Advancing our understanding of these cancers and developing effective strategies for diagnosis. The study will use aminolaevulinic acid (ALA) as a source of protoporphyrin IX (PpIX) to allow the detection of hypoxia signal. More specifically, the oxygen imager gathers the delayed fluorescence (DF) of PpIX, which intensity is inversely proportional to tissue mitochondrial oxygen content. This provides qualitative contrast on hypoxic regions with submillimeter spatial resolution. Transient hypoxia is a clear indicator of tumor tissue. We will validate the combination of hypoxia imaging with palpation as a non-invasive technique to detect cutaneous malignant lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Chapman, MD, Principal Investigator — Dartmouth
Locations (1):
- Dartmouth Hitchcock, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share identifiable data. All data will be owned and maintained by Dartmouth.